CLINICAL TRIAL: NCT00873223
Title: Insulin Detemir Co-administered With Liraglutide: An Open Label Trial to Assess Insulin Detemir and Liraglutide Pharmacokinetics and Pharmacodynamics Following Liraglutide Therapy in Subjects With Type 2 Diabetes
Brief Title: Examination of the Effects of Liraglutide on the Mode of Action of Insulin Detemir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN2211-3673
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: liraglutide; Drug: insulin detemir

INTERVENTIONS:
Drug: liraglutide — Subjects will self-inject liraglutide subcutaneously daily during the trial and three euglycemic clamps will be performed: one without liraglutide (insulin detemir alone), the second with only liraglutide treatment and the third with liraglutide and insulin detemir administration
Drug: insulin detemir — Subjects will self-inject liraglutide subcutaneously daily during the trial and three euglycemic clamps will be performed: one without liraglutide (insulin detemir alone), the second with only liraglutide treatment and the third with liraglutide and insulin detemir administration

SUMMARY:
This trial is conducted in the United States. The aim of this clinical trial is to investigate whether chronic liraglutide administration affects the mode of action (pharmacokinetics) of insulin detemir

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes
* BMI less than 45.0 kg/m2
* Insulin naive
* Currently treated with Oral Anti-Diabetic drugs (OADs) and metformin with a HbA1c between 7.0 and 9.5% or currently treated with metformin only with a HbA1c between 7.0 and 10.0%

Exclusion Criteria:

* Any clinically significant disease other than type 2 diabetes
* Currently using daily insulin
* Thiazolidinione use or other injectable diabetes medications within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Insulin detemir pharmacokinetics with and without liraglutide administration | at approx. 12 weeks (including screening, washout and evaluation period)

SECONDARY OUTCOMES:
Pharmacokinetics of liraglutide with and without insulin detemir | at approx. 12 weeks (including screening, washout and evaluation period)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Chula Vista, California, United States

REFERENCES:
- [Result] Morrow L, Hompesch M, Guthrie H, Chang D, Chatterjee DJ. Co-administration of liraglutide with insulin detemir demonstrates additive pharmacodynamic effects with no pharmacokinetic interaction. Diabetes Obes Metab. 2011 Jan;13(1):75-80. doi: 10.1111/j.1463-1326.2010.01322.x. PMID 21114606
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com